CLINICAL TRIAL: NCT01732458
Title: A Phase IIb, Partially-Blinded, Randomized, Active Comparator-Controlled Study to Evaluate the Pharmacokinetics/Pharmacodynamics, Safety, and Tolerability of Aprepitant in Pediatric Patients for the Prevention of Post Operative Nausea and Vomiting
Brief Title: A Study to Evaluate Aprepitant for the Prevention of Post-Operative Nausea and Vomiting in Children (MK-0869-219)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0869-219; 2011-006006-27 (EudraCT Number)
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Results first posted 2017-09-06 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Post-operative Nausea; Post-operative Vomiting
MeSH Terms: interventions — Aprepitant; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study will be conducted as a partially blinded study. PK samples will not be collected from participants in the control group. To maintain a partial blind, approximately 3 participants randomly selected from each age group in each of the aprepitant treatment groups will not have PK sampling. All participants will remain blinded to the study treatment. The investigator and Sponsor will be blinded to the study medication in participants not providing PK samples. The investigator and Sponsor will remain blinded to the aprepitant dose given to participants from whom PK samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Aprepitant Dose 1: Equivalent to 125 mg in Adults (Experimental): Pediatric participants receive a single dose of apprepitant that is equivalent to 125 mg in adults on Day 1 between 1 and 3 hours prior to expected induction of anesthesia, plus placebo for odansetron administered intravenously (IV) immediately prior to anesthesia.
  Interventions: Drug: Aprepitant; Drug: Placebo to match ondansetron
- Aprepitant Dose 2: Equivalent to 40 mg in Adults (Experimental): Pediatric participants receive a single dose of apprepitant that is equivalent to 40 mg in adults on Day 1 between 1 and 3 hours prior to expected induction of anesthesia, plus placebo for odansetron administered IV immediately prior to anesthesia.
  Interventions: Drug: Aprepitant; Drug: Placebo to match ondansetron
- Aprepitant Dose 3: Equivalent to 10 mg in Adults (Experimental): Pediatric participants receive a single dose of apprepitant that is equivalent to 10 mg in adults Day 1 between 1 and 3 hours prior to expected induction of anesthesia, plus placebo for odansetron administered IV immediately prior to anesthesia.
  Interventions: Drug: Aprepitant; Drug: Placebo to match ondansetron
- Ondansetron (Active Comparator): Pediatric participants in the control regimen are administered ondansetron IV on Day 1 immediately prior to induction of anesthesia plus a matching placebo dose to aprepitant as a single oral dose on Day 1 between 1 and 3 hours prior to expected induction of anesthesia.
  Interventions: Drug: Placebo to Aprepitant; Drug: Ondansetron

INTERVENTIONS:
Drug: Aprepitant — Administered as a single oral dose on Day 1 between 1 and 3 hours prior to expected induction of anesthesia. Aprepitant was supplied in a sachet containing a powder for suspension (PFS) that was reconstituted up to total volume of 5 mL using potable water.
  Other Names: MK-0869; EMEND™
  Arms: Aprepitant Dose 1: Equivalent to 125 mg in Adults; Aprepitant Dose 2: Equivalent to 40 mg in Adults; Aprepitant Dose 3: Equivalent to 10 mg in Adults
Drug: Placebo to Aprepitant
  Other Names: Matching placebo to aprepritant was administered as a single oral dose on Day 1 between 1 and 3 hours prior to expected induction of anesthesia.
  Arms: Ondansetron
Drug: Ondansetron — Administered IV at a dose of 4 mg for participants >40 kg in weight and 0.1 mg/kg for participants ≤40 kg in weight. In participants <1 month of age, the dose of ondansetron was administered per the product label or based on local standard of care. Ondansetron was supplied by the Sponsor as vials or ampules, depending on the country.
  Other Names: Zofran
  Arms: Ondansetron
Drug: Placebo to match ondansetron — Participants in the aprepitant regimen received normal saline IV (provided by the site) as the placebo for ondansetron on Day 1, immediately prior to induction of anesthesia.
  Arms: Aprepitant Dose 1: Equivalent to 125 mg in Adults; Aprepitant Dose 2: Equivalent to 40 mg in Adults; Aprepitant Dose 3: Equivalent to 10 mg in Adults

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK), safety, and tolerability of aprepitant for the prevention of post-operative nausea and vomiting (PONV) in pediatric participants.

Post-operative aprepitant plasma concentrations will be evaluated with a non-compartmental analysis (NCA) at each dose and for each age cohort. Full PK profiles analyzed using population PK modeling and simulation will be described in a separate report.

DETAILED DESCRIPTION:
Because the opportunity to collect specimens for PK analyses in children will be limited, a flexible sparse sampling scheme using ranges of collection times will be utilized which will limit the burden to participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant enrolled at birth should be at least 37 weeks gestation and ≥3 kg of weight
* Scheduled to receive general anesthesia AND must have at least one of the following risk factors for post-operative nausea and vomiting (PONV) in addition to receiving general anesthesia:

  1. scheduled to have a surgery with an associated risk of PONV: tonsillectomy, adenoidectomy, strabismus surgery, dental surgery, hydrocelectomy, orchidopexy or herniorraphy; OR
  2. scheduled to have an operative procedure associated with PONV: intraoperative opioid use or anticipated opioid administration within the first 24 hours following surgery.

Exclusion Criteria:

* Emergency surgery for a life-threatening condition
* Scheduled to receive propofol for maintenance of anesthesia (Note: propofol is permitted for induction of anesthesia).
* Expected to receive opioid antagonists (e.g., naloxone, naltrexone) or

benzodiazepine antagonists (e.g., flumazenil)

* Scheduled to undergo cardiac or neurosurgery
* Vomiting caused by any organic etiology (such as gastric outlet

obstruction or small bowel obstruction)

* Vomiting within 24 hours prior to surgery
* Participant had a nasogastric or oral gastric tube intra- or post-operatively for suctioning gastric contents (note: nasogastric or oral gastric tube intra- or post-operatively could only be used for feeding. Participants were to be excluded if a nasogastric or oral gastric tube for suctioning was routinely used for the type of surgery being performed)
* Active infection (e.g., pneumonia), congestive heart failure, bradyarrythmia, any uncontrolled disease (e.g., diabetic ketoacidosis, gastrointestinal obstruction) except for malignancy, or a history of any illness which in the opinion of the investigator, might confound the results of the study or pose unwarranted risk to the participant
* Use of any illicit drugs, including marijuana or has current evidence of alcohol abuse

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 229 (Actual)
Dates: Start 2013-02-12 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Salman FT, DiCristina C, Chain A, Afzal AS. Pharmacokinetics and pharmacodynamics of aprepitant for the prevention of postoperative nausea and vomiting in pediatric subjects. J Pediatr Surg. 2019 Jul;54(7):1384-1390. doi: 10.1016/j.jpedsurg.2018.09.006. Epub 2018 Sep 21. PMID 30381138

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 262 screened for inclusion, 229 were randomized to treatment. 1 participant was inadvertently randomized to a 2.5 mg aprepitant dose arm that was not evaluated in this study; therefore the participant was not included in any analyses. Of remaining 228 randomized participants, 8 did not receive treatment.
Groups:
- Aprepitant Dose 1: Equivalent to 125 mg in Adults: Pediatric participants received a single dose of apprepitant that was equivalent to 125 mg in adults on Day 1 between 1 and 3 hours prior to expected induction of anesthesia, plus placebo for odansetron administered intravenously (IV) immediately prior to anesthesia.
- Aprepitant Dose 2: Equivalent to 40 mg in Adults: Pediatric participants received a single dose of apprepitant that was equivalent to 40 mg in adults on Day 1 between 1 and 3 hours prior to expected induction of anesthesia, plus placebo for odansetron administered IV immediately prior to anesthesia.
- Aprepitant Dose 3: Equivalent to 10 mg in Adults: Pediatric participants received a single dose of apprepitant that was equivalent to 10 mg in adults Day 1 between 1 and 3 hours prior to expected induction of anesthesia, plus placebo for odansetron administered IV immediately prior to anesthesia.
- Ondansetron: Pediatric participants in the control regimen were administered ondansetron IV on Day 1 immediately prior to induction of anesthesia plus a matching placebo dose to aprepitant as a single oral dose on Day 1 between 1 and 3 hours prior to expected induction of anesthesia.
Period: Overall Study
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults | Aprepitant Dose 2: Equivalent to 40 mg in Adults | Aprepitant Dose 3: Equivalent to 10 mg in Adults | Ondansetron
Started | 60 | 58 | 58 | 52
Treated | 57 | 55 | 56 | 52
Completed | 57 | 53 | 55 | 50
Not Completed | 3 | 5 | 3 | 2
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — Non-Compliance With Study Drug | 0 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 2 | 2 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 2
Not completed — Screen Failure | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Participants as Treated (APaT) population; all randomized participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults | Aprepitant Dose 2: Equivalent to 40 mg in Adults | Aprepitant Dose 3: Equivalent to 10 mg in Adults | Ondansetron | Total
Number analyzed (Participants) | 57 | 55 | 56 | 52 | 220
Age, Continuous [Mean (Standard Deviation); unit: months] | 90.4 (64.3) | 87.5 (64.6) | 85.1 (59.7) | 86.0 (65.0) | 87.3 (63.0)
Age, Customized [Number; unit: participants]
  Birth to <2 years | 14 | 12 | 13 | 11 | 50
  2 years to <6 years | 14 | 14 | 15 | 14 | 57
  6 years to <12 years | 13 | 15 | 14 | 13 | 55
  12 years to 17 years | 16 | 14 | 14 | 14 | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 28 | 16 | 86
  Male | 34 | 36 | 28 | 36 | 134

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Aprepitant From Time 0 to the Last Measurable Concentration (AUC0-last) Following Administration of 125 mg Dose Equivalent in 12 to 17 Year Age Group
Description: AUC0-last was analyzed independently for participants in the 125 mg dose equivalent arm aged 12 to 17 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant AUC0-last assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma AUC0-last was evaluated using a noncompartmental analysis (NCA). The limit of quantitation (LOQ) value for this analysis was 10 ng/mL.
Time Frame: 30-60 minutes pre-administration, 2-4 hours post administration, 5-7 hours post administration, 8-10 hours post administration
Population: Participants aged 12 to 17 years who received a single dose of 125 mg aprepitant prior to surgery with available plasma samples were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Aprepitant Dose 1: Equivalent to 125 mg in Adults; 12 to 17: Subset of pediatric participants receiving a single dose of oral aprepitant approximating adult equivalent dose of 125 mg on Day 1 between 1 and 3 hours prior to expected induction of anesthesia that were aged 12 to 17 years old.
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults; 12 to 17
Number analyzed (Participants) | 10
hr*ng/mL | 7120 (33.0)

2. Primary Outcome: Maximum Concentration (Cmax) of Aprepitant Following Administration of 125 mg Dose Equivalent in 12 to 17 Year Age Group
Description: Cmax was analyzed independently for participants in the 125 mg dose equivalent arm aged 12 to 17 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Cmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Cmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults; 12 to 17
Number analyzed (Participants) | 10
ng/mL | 1340 (43.9)

3. Primary Outcome: Time to Maximum Concentration (Tmax) of Aprepitant Following Administration of 125 mg Dose Equivalent in 12 to 17 Year Age Group
Description: Tmax was analyzed independently for participants in the 125 mg dose equivalent arm aged 12 to 17 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Tmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Tmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (hr)
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults; 12 to 17
Number analyzed (Participants) | 10
hour (hr) | 4.86 (56.5)

4. Primary Outcome: AUC0-last of Aprepitant Following Administration of 125 mg Dose Equivalent in 6 to <12 Year Age Group
Description: AUC0-last was analyzed independently for participants in the 125 mg dose equivalent arm aged 6 to <12 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant AUC0-last assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma AUC0-last was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: Participants aged 6 to <12 years who received a single dose of 125 mg aprepitant prior to surgery with available plasma samples were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Aprepitant Dose 1: Equivalent to 125 mg in Adults; 6 to <12: Subset of pediatric participants receiving a single dose of oral aprepitant approximating adult equivalent dose of 125 mg on Day 1 between 1 and 3 hours prior to expected induction of anesthesia that were aged 6 to <12 years old.
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults; 6 to <12
Number analyzed (Participants) | 11
hr*ng/mL | 10300 (39.5)

5. Primary Outcome: Cmax of Aprepitant Following Administration of 125 mg Dose Equivalent in 6 to <12 Year Age Group
Description: Cmax was analyzed independently for participants in the 125 mg dose equivalent arm aged 6 to <12 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Cmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Cmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults; 6 to <12
Number analyzed (Participants) | 11
ng/mL | 1870 (53.0)

6. Primary Outcome: Tmax of Aprepitant Following Administration of 125 mg Dose Equivalent in 6 to <12 Year Age Group
Description: Tmax was analyzed independently for participants in the 125 mg dose equivalent arm aged 6 to <12 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Tmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Tmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults; 6 to <12
Number analyzed (Participants) | 11
hr | 6.82 (26.8)

7. Primary Outcome: AUC0-last of Aprepitant Following Administration of 125 mg Dose Equivalent in 2 to <6 Year Age Group
Description: AUC0-last was analyzed independently for participants in the 125 mg dose equivalent arm aged 2 to <6 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant AUC0-last assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma AUC0-last was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: Participants aged 2 to <6 years who received a single dose of 125 mg aprepitant prior to surgery with available plasma samples were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Aprepitant Dose 1: Equivalent to 125 mg in Adults; 2 to <6: Subset of pediatric participants receiving a single dose of oral aprepitant approximating adult equivalent dose of 125 mg on Day 1 between 1 and 3 hours prior to expected induction of anesthesia that were aged 2 to <6 years old.
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults; 2 to <6
Number analyzed (Participants) | 10
hr*ng/mL | 12000 (39.7)

8. Primary Outcome: Cmax of Aprepitant Following Administration of 125 mg Dose Equivalent in 2 to <6 Year Age Group
Description: Cmax was analyzed independently for participants in the 125 mg dose equivalent arm aged 2 to <6 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Cmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Cmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults; 2 to <6
Number analyzed (Participants) | 10
ng/mL | 2260 (35.7)

9. Primary Outcome: Tmax of Aprepitant Following Administration of 125 mg Dose Equivalent in 2 to <6 Year Age Group
Description: Tmax was analyzed independently for participants in the 125 mg dose equivalent arm aged 2 to <6 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Tmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Tmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults; 2 to <6
Number analyzed (Participants) | 10
hr | 4.91 (51.9)

10. Primary Outcome: AUC0-last of Aprepitant Following Administration of 125 mg Dose Equivalent in Birth to <2 Year Age Group
Description: AUC0-last was analyzed independently for participants in the 125 mg dose equivalent arm aged birth to <2 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant AUC0-last assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma AUC0-last was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: Participants aged birth to <2 years who received a single dose of 125 mg aprepitant prior to surgery with available plasma samples were analyzed. Two participants were excluded from the analysis, due to a missing 8-hour post-dose sample and aprepitant concentration in the pre-dose sample, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Aprepitant Dose 1: Equivalent to 125 mg in Adults; Birth to <2: Subset of pediatric participants receiving a single dose of oral aprepitant approximating adult equivalent dose of 125 mg on Day 1 between 1 and 3 hours prior to expected induction of anesthesia that were aged birth to <2 years old.
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults; Birth to <2
Number analyzed (Participants) | 8
hr*ng/mL | 6410 (67.8)

11. Primary Outcome: Cmax of Aprepitant Following Administration of 125 mg Dose Equivalent in Birth to <2 Year Age Group
Description: Cmax was analyzed independently for participants in the 125 mg dose equivalent arm aged birth to <2 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Cmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative plasma Cmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: Participants aged birth to <2 years who received a single dose of 125 mg aprepitant prior to surgery with available plasma samples were analyzed. One participant was excluded from the analysis due to aprepitant concentration in the pre-dose sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults; Birth to <2
Number analyzed (Participants) | 9
ng/mL | 1280 (78.5)

12. Primary Outcome: Tmax of Aprepitant Following Administration of 125 mg Dose Equivalent in Birth to <2 Year Age Group
Description: Tmax was analyzed independently for participants in the 125 mg dose equivalent arm aged birth to <2 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Tmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Tmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: Participants aged birth to <2 years who received a single dose of 125 mg aprepitant prior to surgery with available plasma samples were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults; Birth to <2
Number analyzed (Participants) | 10
hr | 4.71 (51.3)

13. Primary Outcome: AUC0-last Following Administration of 40 mg Dose Equivalent in 12 to 17 Year Age Group
Description: AUC0-last was analyzed independently for participants in the 40 mg dose equivalent arm aged 12 to 17 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant AUC0-last assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma AUC0-last was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: Participants aged 12 to 17 years who received a single dose of 40 mg aprepitant prior to surgery with available plasma samples were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Aprepitant Dose 2: Equivalent to 40 mg in Adults; 12 to 17: Subset of pediatric participants receiving a single dose of oral aprepitant approximating adult equivalent dose of 40 mg on Day 1 between 1 and 3 hours prior to expected induction of anesthesia that were aged 12 to 17 years old.
Arm/Group | Aprepitant Dose 2: Equivalent to 40 mg in Adults; 12 to 17
Number analyzed (Participants) | 11
hr*ng/mL | 2570 (41.5)

14. Primary Outcome: Cmax Following Administration of 40 mg Dose Equivalent in 12 to 17 Year Age Group
Description: Cmax was analyzed independently for participants in the 40 mg dose equivalent arm aged 12 to 17 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Cmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Cmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Aprepitant Dose 2: Equivalent to 40 mg in Adults; 12 to 17
Number analyzed (Participants) | 11
ng/mL | 513 (41.6)

15. Primary Outcome: Tmax Following Administration of 40 mg Dose Equivalent in 12 to 17 Year Age Group
Description: Tmax was analyzed independently for participants in the 40 mg dose equivalent arm aged 12 to 17 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Tmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Tmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Aprepitant Dose 2: Equivalent to 40 mg in Adults; 12 to 17
Number analyzed (Participants) | 11
hr | 4.17 (69.4)

16. Primary Outcome: AUC0-last of Aprepitant Following Administration of 40 mg Dose Equivalent in 6 to <12 Year Age Group
Description: AUC0-last was analyzed independently for participants in the 40 mg dose equivalent arm aged 6 to <12 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant AUC0-last assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma AUC0-last was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: Participants aged 6 to <12 years who received a single dose of 40 mg aprepitant prior to surgery with available plasma samples were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Aprepitant Dose 2: Equivalent to 40 mg in Adults; 6 to <12: Subset of pediatric participants receiving a single dose of oral aprepitant approximating adult equivalent dose of 40 mg on Day 1 between 1 and 3 hours prior to expected induction of anesthesia that were aged 6 to <12 years old.
Arm/Group | Aprepitant Dose 2: Equivalent to 40 mg in Adults; 6 to <12
Number analyzed (Participants) | 11
hr*ng/mL | 4730 (60.7)

17. Primary Outcome: Cmax of Aprepitant Following Administration of 40 mg Dose Equivalent in 6 to <12 Year Age Group
Description: Cmax was analyzed independently for participants in the 40 mg dose equivalent arm aged 6 to <12 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Cmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Cmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Aprepitant Dose 2: Equivalent to 40 mg in Adults; 6 to <12
Number analyzed (Participants) | 11
ng/mL | 930 (66.7)

18. Primary Outcome: Tmax of Aprepitant Following Administration of 40 mg Dose Equivalent in 6 to <12 Year Age Group
Description: Tmax was analyzed independently for participants in the 40 mg dose equivalent arm aged 6 to <12 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Tmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Tmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Aprepitant Dose 2: Equivalent to 40 mg in Adults; 6 to <12
Number analyzed (Participants) | 11
hr | 4.22 (53.4)

19. Primary Outcome: AUC0-last of Aprepitant Following Administration of 40 mg Dose Equivalent in 2 to <6 Year Age Group
Description: AUC0-last was analyzed independently for participants in the 40 mg dose equivalent arm aged 2 to <6 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant AUC0-last assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma AUC0-last was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: Participants aged 2 to <6 years who received a single dose of 40 mg aprepitant prior to surgery with available plasma samples were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Aprepitant Dose 2: Equivalent to 40 mg in Adults; 2 to <6: Subset of pediatric participants receiving a single dose of oral aprepitant approximating adult equivalent dose of 40 mg on Day 1 between 1 and 3 hours prior to expected induction of anesthesia that were aged 2 to <6 years old.
Arm/Group | Aprepitant Dose 2: Equivalent to 40 mg in Adults; 2 to <6
Number analyzed (Participants) | 9
hr*ng/mL | 6320 (78.1)

20. Primary Outcome: Cmax of Aprepitant Following Administration of 40 mg Dose Equivalent in 2 to <6 Year Age Group
Description: Cmax was analyzed independently for participants in the 40 mg dose equivalent arm aged 2 to <6 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Cmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Cmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Aprepitant Dose 2: Equivalent to 40 mg in Adults; 2 to <6
Number analyzed (Participants) | 9
ng/mL | 1290 (81.7)

21. Primary Outcome: Tmax of Aprepitant Following Administration of 40 mg Dose Equivalent in 2 to <6 Year Age Group
Description: Tmax was analyzed independently for participants in the 40 mg dose equivalent arm aged 2 to <6 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Tmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Tmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Aprepitant Dose 2: Equivalent to 40 mg in Adults; 2 to <6
Number analyzed (Participants) | 9
hr | 3.35 (43.0)

22. Primary Outcome: AUC0-last of Aprepitant Following Administration of 40 mg Dose Equivalent in Birth to <2 Year Age Group
Description: AUC0-last was analyzed independently for participants in the 40 mg dose equivalent arm aged birth to <2 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant AUC0-last assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma AUC0-last was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: Participants aged birth to <2 years who received a single dose of 40 mg aprepitant prior to surgery with available plasma samples were analyzed. One participant was excluded from the analysis due aprepitant concentration in the pre-dose sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Aprepitant Dose 2: Equivalent to 40 mg in Adults; Birth to <2: Subset of pediatric participants receiving a single dose of oral aprepitant approximating adult equivalent dose of 40 mg on Day 1 between 1 and 3 hours prior to expected induction of anesthesia that were aged birth to <2 years old.
Arm/Group | Aprepitant Dose 2: Equivalent to 40 mg in Adults; Birth to <2
Number analyzed (Participants) | 6
hr*ng/mL | 7910 (153.2)

23. Primary Outcome: Cmax of Aprepitant Following Administration of 40 mg Dose Equivalent in Birth to <2 Year Age Group
Description: Cmax was analyzed independently for participants in the 40 mg dose equivalent arm aged birth to <2 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Cmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Cmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Aprepitant Dose 2: Equivalent to 40 mg in Adults; Birth to <2
Number analyzed (Participants) | 6
ng/mL | 1570 (146.3)

24. Primary Outcome: Tmax of Aprepitant Following Administration of 40 mg Dose Equivalent in Birth to <2 Year Age Group
Description: Tmax was analyzed independently for participants in the 40 mg dose equivalent arm aged birth to <2 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Tmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Tmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: Participants aged birth to <2 years who received a single dose of 40 mg aprepitant prior to surgery with available plasma samples were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Aprepitant Dose 2: Equivalent to 40 mg in Adults; Birth to <2
Number analyzed (Participants) | 7
hr | 4.94 (38.0)

25. Primary Outcome: AUC0-last Following Administration of 10 mg Dose Equivalent in 12 to 17 Year Age Group
Description: AUC0-last was analyzed independently for participants in the 10 mg dose equivalent arm aged 12 to 17 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant AUC0-last assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma AUC0-last was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: Participants aged 12 to 17 years who received a single dose of 10 mg aprepitant prior to surgery with available plasma samples were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Aprepitant Dose 3: Equivalent to 10 mg in Adults; 12 to 17: Subset of pediatric participants receiving a single dose of oral aprepitant approximating adult equivalent dose of 10 mg on Day 1 between 1 and 3 hours prior to expected induction of anesthesia that were aged 12 to 17 years old.
Arm/Group | Aprepitant Dose 3: Equivalent to 10 mg in Adults; 12 to 17
Number analyzed (Participants) | 10
hr*ng/mL | 806 (51.9)

26. Primary Outcome: Cmax of Aprepitant Following Administration of 10 mg Dose Equivalent in 12 to 17 Year Age Group
Description: Cmax was analyzed independently for participants in the 10 mg dose equivalent arm aged 12 to 17 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Cmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Cmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Aprepitant Dose 3: Equivalent to 10 mg in Adults; 12 to 17
Number analyzed (Participants) | 10
ng/mL | 131 (50.8)

27. Primary Outcome: Tmax of Aprepitant Following Administration of 10 mg Dose Equivalent in 12 to 17 Year Age Group
Description: Tmax was analyzed independently for participants in the 10 mg dose equivalent arm aged 12 to 17 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Tmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Tmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Aprepitant Dose 3: Equivalent to 10 mg in Adults; 12 to 17
Number analyzed (Participants) | 10
hr | 3.53 (54.1)

28. Primary Outcome: AUC0-last of Aprepitant Following Administration of 10 mg Dose Equivalent in 6 to <12 Year Age Group
Description: AUC0-last was analyzed independently for participants in the 10 mg dose equivalent arm aged 6 to <12 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant AUC0-last assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma AUC0-last was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: Participants aged 6 to <12 years who received a single dose of 10 mg aprepitant prior to surgery with available plasma samples were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Aprepitant Dose 3: Equivalent to 10 mg in Adults; 6 to <12: Subset of pediatric participants receiving a single dose of oral aprepitant approximating adult equivalent dose of 10 mg on Day 1 between 1 and 3 hours prior to expected induction of anesthesia that were aged 6 to <12 years old.
Arm/Group | Aprepitant Dose 3: Equivalent to 10 mg in Adults; 6 to <12
Number analyzed (Participants) | 10
hr*ng/mL | 1390 (77.0)

29. Primary Outcome: Cmax of Aprepitant Following Administration of 10 mg Dose Equivalent in 6 to <12 Year Age Group
Description: Cmax was analyzed independently for participants in the 10 mg dose equivalent arm aged 6 to <12 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Cmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Cmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Aprepitant Dose 3: Equivalent to 10 mg in Adults; 6 to <12
Number analyzed (Participants) | 10
ng/mL | 289 (128.4)

30. Primary Outcome: Tmax of Aprepitant Following Administration of 10 mg Dose Equivalent in 6 to <12 Year Age Group
Description: Tmax was analyzed independently for participants in the 10 mg dose equivalent arm aged 6 to <12 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Tmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Tmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Aprepitant Dose 3: Equivalent to 10 mg in Adults; 6 to <12
Number analyzed (Participants) | 10
hr | 3.75 (57.9)

31. Primary Outcome: AUC0-last of Aprepitant Following Administration of 10 mg Dose Equivalent in 2 to <6 Year Age Group
Description: AUC0-last was analyzed independently for participants in the 10 mg dose equivalent arm aged 2 to <6 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant AUC0-last assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma AUC0-last was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: Participants aged 2 to <6 years who received a single dose of 10 mg aprepitant prior to surgery with available plasma samples were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Aprepitant Dose 3: Equivalent to 10 mg in Adults; 2 to <6: Subset of pediatric participants receiving a single dose of oral aprepitant approximating adult equivalent dose of 10 mg on Day 1 between 1 and 3 hours prior to expected induction of anesthesia that were aged 2 to <6 years old.
Arm/Group | Aprepitant Dose 3: Equivalent to 10 mg in Adults; 2 to <6
Number analyzed (Participants) | 10
hr*ng/mL | 1580 (45.2)

32. Primary Outcome: Cmax of Aprepitant Following Administration of 10 mg Dose Equivalent in 2 to <6 Year Age Group
Description: Cmax was analyzed independently for participants in the 10 mg dose equivalent arm aged 2 to <6 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Cmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Cmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 31
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Aprepitant Dose 3: Equivalent to 10 mg in Adults; 2 to <6
Number analyzed (Participants) | 10
ng/mL | 300 (49.9)

33. Primary Outcome: Tmax of Aprepitant Following Administration of 10 mg Dose Equivalent in 2 to <6 Year Age Group
Description: Tmax was analyzed independently for participants in the 10 mg dose equivalent arm aged 2 to <6 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Tmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Tmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 31
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Aprepitant Dose 3: Equivalent to 10 mg in Adults; 2 to <6
Number analyzed (Participants) | 10
hr | 3.36 (45.8)

34. Primary Outcome: AUC0-last of Aprepitant Following Administration of 10 mg Dose Equivalent in Birth to <2 Year Age Group
Description: AUC0-last was analyzed independently for participants in the 10 mg dose equivalent arm aged from birth to <2 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant AUC0-last assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma AUC0-last was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: Participants aged birth to <2 years who received a single dose of 10 mg aprepitant prior to surgery with available plasma samples were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Aprepitant Dose 3: Equivalent to 10 mg in Adults; Birth to <2: Subset of pediatric participants receiving a single dose of oral aprepitant approximating adult equivalent dose of 40 mg on Day 1 between 1 and 3 hours prior to expected induction of anesthesia that were aged birth to <2 years old.
Arm/Group | Aprepitant Dose 3: Equivalent to 10 mg in Adults; Birth to <2
Number analyzed (Participants) | 10
hr*ng/mL | 1800 (107.8)

35. Primary Outcome: Cmax of Aprepitant Following Administration of 10 mg Dose Equivalent in Birth to <2 Year Age Group
Description: Cmax was analyzed independently for participants in the 10 mg dose equivalent arm aged from birth to <2 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Cmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Cmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Aprepitant Dose 3: Equivalent to 10 mg in Adults; Birth to <2
Number analyzed (Participants) | 10
ng/mL | 336 (112.0)

36. Primary Outcome: Tmax of Aprepitant Following Administration of 10 mg Dose Equivalent in Birth to <2 Year Age Group
Description: Tmax was analyzed independently for participants in the 10 mg dose equivalent arm aged from birth to <2 years old due to age- and dose-dependent differences in aprepitant absorption and clearance. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. Plasma for aprepitant Tmax assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Post-operative aprepitant plasma Tmax was evaluated using an NCA. The LOQ value for this analysis was 10 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Aprepitant Dose 3: Equivalent to 10 mg in Adults; Birth to <2
Number analyzed (Participants) | 10
hr | 4.11 (48.2)

37. Primary Outcome: Area Under the Concentration-time Curve of Aprepitant From Time 0 to Infinity (AUC0-inf) Following Administration of Single Dose
Description: Plasma for aprepitant AUC0-inf assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. AUC0-inf data were to be log transformed and analyzed via a linear mixed-effects model containing fixed effects for age for each dose level tested.
Time Frame: as for outcome 1
Population: Due to the lack of samples beyond 8 hours after dose, the assessment of the terminal elimination phase of the PK profiles was limited and derivation of parameters dependent on lambda (e.g. AUC0-inf) was not possible.
Groups:
- Aprepitant Dose 1: Equivalent to 125 mg in Adults: Pediatric participants received a single dose of apprepitant that was equivalent to 125 mg in adults on Day 1 between 1 and 3 hours prior to expected induction of anesthesia, plus placebo for odansetron administered IV immediately prior to anesthesia.
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults | Aprepitant Dose 2: Equivalent to 40 mg in Adults | Aprepitant Dose 3: Equivalent to 10 mg in Adults | Ondansetron
Number analyzed (Participants) | 0 | 0 | 0 | 0

38. Primary Outcome: Apparent Total Clearance (CL/F) of Aprepitant From Plasma Following Administration of Single Dose
Description: Plasma for aprepitant CL/F assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. CL/F data were to be log transformed and analyzed via a linear mixed-effects model containing fixed effects for age for each dose level tested.
Time Frame: as for outcome 1
Population: Due to the lack of samples beyond 8 hours after dose, the assessment of the terminal elimination phase of the PK profiles was limited and derivation of parameters dependent on lambda (e.g. CL/F) was not possible.
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults | Aprepitant Dose 2: Equivalent to 40 mg in Adults | Aprepitant Dose 3: Equivalent to 10 mg in Adults | Ondansetron
Number analyzed (Participants) | 0 | 0 | 0 | 0

39. Primary Outcome: Apparent Terminal Half-life (t ½) of Aprepitant Following Administration of Single Dose
Description: Plasma for aprepitant t ½ assessment was obtained at 30-60 minutes prior to aprepitant administration, 2-4 hours post aprepitant administration, 5-7 hours post aprepitant administration, and 8-10 hours post aprepitant administration. Because the opportunity to collect specimens for PK analyses in children is limited, a flexible sparse sampling scheme using ranges of collection times was to be utilized which would limit the burden to participants. t ½ data were to be log transformed and analyzed via a linear mixed-effects model containing fixed effects for age for each dose level tested.
Time Frame: as for outcome 1
Population: Due to the lack of samples beyond 8 hours after dose, the assessment of the terminal elimination phase of the PK profiles was limited and derivation of parameters dependent on lambda (e.g. t ½) was not possible.
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults | Aprepitant Dose 2: Equivalent to 40 mg in Adults | Aprepitant Dose 3: Equivalent to 10 mg in Adults | Ondansetron
Number analyzed (Participants) | 0 | 0 | 0 | 0

40. Primary Outcome: Percentage of Participants Experiencing at Least One Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening of a pre-existing condition which is temporally associated with the use of the SPONSOR's product, was also an AE. Changes resulting from normal growth and development which did not vary significantly in frequency or severity from expected levels were not to be considered adverse events. Vomiting and retching were not defined as AEs during the period of data collection (24 hours following the end of surgery) unless they met the definition of an SAE. The percentage of participants experiencing ≥1 AE was reported by dose group.
Time Frame: From pre-operative phase up to Follow-up (Day 1 to Day 15)
Population: All randomized participants who received at least one dose of study treatment were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults | Aprepitant Dose 2: Equivalent to 40 mg in Adults | Aprepitant Dose 3: Equivalent to 10 mg in Adults | Ondansetron
Number analyzed (Participants) | 57 | 55 | 56 | 52
percentage of participants | 31.6 | 43.6 | 35.7 | 48.1
Statistical Analysis 1: Comparison: Aprepitant Dose 1: Equivalent to 125 mg in Adults vs Ondansetron; The Miettinen and Nurminen method was used to provide 95% confidence intervals (CIs) for between-treatment differences in the percentage of participants with events; Test type: Superiority or Other; Difference in Percentage vs. Ondansetron = -16.5, 95% CI 2-sided [-34.0 to 2.0]
Statistical Analysis 2: Comparison: Aprepitant Dose 2: Equivalent to 40 mg in Adults vs Ondansetron; [analysis description as in outcome 40, analysis 1]; Test type: Superiority or Other; Difference in Percentage vs. Ondansetron = -4.4, 95% CI 2-sided [-22.9 to 14.3]
Statistical Analysis 3: Comparison: Aprepitant Dose 3: Equivalent to 10 mg in Adults vs Ondansetron; [analysis description as in outcome 40, analysis 1]; Test type: Superiority or Other; Difference in Percentage vs. Ondansetron = -12.4, 95% CI 2-sided [-30.3 to 6.3]

41. Primary Outcome: Percentage of Participants Discontinuing Study Due to an AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening of a pre-existing condition which is temporally associated with the use of the SPONSOR's product, was also an AE. Changes resulting from normal growth and development which did not vary significantly in frequency or severity from expected levels were not to be considered adverse events. Vomiting and retching were not defined as AEs during the period of data collection (24 hours following the end of surgery) unless they met the definition of an SAE. The percentage of participants discontinuing study due to an AE was reported by dose group.
Time Frame: From pre-operative phase up to Follow-up (Day 1 to Day 15)
Population: All randomized participants who received at least one dose of study treatment were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Aprepitant Dose 1: Equivalent to 125 mg in Adults | Aprepitant Dose 2: Equivalent to 40 mg in Adults | Aprepitant Dose 3: Equivalent to 10 mg in Adults | Ondansetron
Number analyzed (Participants) | 57 | 55 | 56 | 52
percentage of participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From pre-operative phase up to Follow-up (up to 17 days)
Description: All randomized participants who received at least one dose of study treatment were analyzed (N=220). 1 participant was inadvertently randomized to a 2.5 mg aprepitant dose group which was not assessed for overall efficacy and safety, thus participant was not included in this safety analysis.
Groups:
- Aprepitant 125 mg Adult Equivalent (Dose 1): Pediatric participants received a single dose of apprepitant that was equivalent to 125 mg in adults on Day 1 between 1 and 3 hours prior to expected induction of anesthesia, plus placebo for odansetron administered IV immediately prior to anesthesia.
- Aprepitant 40 mg Adult Equivalent (Dose 2): Pediatric participants received a single dose of apprepitant that was equivalent to 40 mg in adults on Day 1 between 1 and 3 hours prior to expected induction of anesthesia, plus placebo for odansetron administered IV immediately prior to anesthesia.
- Aprepitant 10 mg Adult Equivalent (Dose 3): Pediatric participants received a single dose of apprepitant that was equivalent to 10 mg in adults Day 1 between 1 and 3 hours prior to expected induction of anesthesia, plus placebo for odansetron administered IV immediately prior to anesthesia.
Arm/Group | Aprepitant 125 mg Adult Equivalent (Dose 1) | Aprepitant 40 mg Adult Equivalent (Dose 2) | Aprepitant 10 mg Adult Equivalent (Dose 3) | Ondansetron
Serious Adverse Events (participants affected / at risk) | 0/57 | 6/55 | 1/56 | 2/52
Other Adverse Events (participants affected / at risk) | 11/57 | 11/55 | 12/56 | 16/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant 125 mg Adult Equivalent (Dose 1) (N=57) | Aprepitant 40 mg Adult Equivalent (Dose 2) (N=55) | Aprepitant 10 mg Adult Equivalent (Dose 3) (N=56) | Ondansetron (N=52)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Male genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant 125 mg Adult Equivalent (Dose 1) (N=57) | Aprepitant 40 mg Adult Equivalent (Dose 2) (N=55) | Aprepitant 10 mg Adult Equivalent (Dose 3) (N=56) | Ondansetron (N=52)
Abdominal pain (Gastrointestinal disorders) | 3 (6) | 3 (4) | 4 (6) | 4 (6)
Vomiting (Gastrointestinal disorders) | 2 (3) | 3 (3) | 2 (3) | 4 (6)
Pyrexia (General disorders) | 3 (5) | 1 (1) | 3 (5) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 4 (8) | 4 (4) | 3 (3) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.